CLINICAL TRIAL: NCT06011629
Title: Prospective Evaluation of Type IV Hypersensitivity Reactions After Aquacel Dressing Application in Partial and Total Joint Arthroplasty Patients
Brief Title: Aquacel Hypersensitivity Dressing in TJAs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Vasili Karas, Assistant Professor, Orthopaedic Surgery Adult Reconstruction and Replacement, Rush University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23050308
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Contact Allergic Dermatitis; Adverse Skin Reaction
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arthroplasty-naïve Aquacel group (Other): All subject's receive the same dressing, this group is comprised of patients consented to the study and will receive the Aquacel dressing but have not had previous joint replacement surgery. Therefore, we consider them the arthroplasty-naïve Aquacel group.
  Interventions: Device: Aquacel dressing
- Prior Aquacel group (Other): All subject's receive the Aquacel dressing, this group is comprised of patients who have undergone previous joint replacement surgery (hip or knee) and have had a Aquacel dressing. This also includes patients who have had prior exposure to glue/mesh dressing either as a patient or healthcare worker.
  Interventions: Device: Aquacel dressing

INTERVENTIONS:
Device: Aquacel dressing — Patients will be recruited into the study after completing a standard questionnaire for pre-operative enrollment. After meeting inclusion criteria and passing the screening process, the patient will be enrolled into the study. Arthroplasty-naïve patients will be compared to prior total joint arthroplasty patients who received a Aquacel dressing postoperatively.

SUMMARY:
The aim of this multi-surgeon, single institution study is to prospectively evaluate the incidence of allergic contact dermatitis (ACD) following application of AQUACEL Ag, a silver-containing hydrofiber dressing, in total hip and knee arthroplasty patients. Arthroplasty-naïve patients will be compared to prior total joint arthroplasty patients who received a Aquacel dressing postoperatively.

DETAILED DESCRIPTION:
Level I: Prospective Cohort Study Patients will be recruited into the study after completing a standard questionnaire for pre-operative enrollment. After meeting inclusion criteria and passing the screening process, the patient will be enrolled into the study. Variables of interest related to sociodemographic status, operative details and postoperative outcomes.

Sample Size:

A power analysis to determine how many patients need to be enrolled was performed with a rate of ACD in the AQUACEL Ag naïve group and the AQAUCEL Ag-exposed group of 1% and 2%, respectively. A one-tailed z-test of proportions between the two groups with 80% power, a 5% level of significance, and 1:1 allocation ratio, requires a sample size of 314 (157 per group). To account for 20% attrition rate amongst both cohorts, we plan to enroll 400 patients (200 each group).

Demographic/Patient Specific Data Collected:

Age, Sex, Body Mass Index (BMI), Allergy History, Past Surgical History, Prior exposure to surgical dressing (Either occupational (i.e. healthcare worker) or as a patient), Number of prior arthroplasty surgeries with AQUACEL Ag dressing (i.e. 0, 1, 2, 3), Past adverse reaction to AQUACEL Ag dressing, Any Adverse Skin Reactions with any past adhesive exposure

Operative details:

Surgical date, Operation/Laterality (THA/TKA/UKA, Left/Right), Length of incision, Patient reported skin check at 1 week (via picture from patient if wound issue/skin reaction present), Size of Rash if present, Provider skin Check at 1st post-operative appointment (2-4 weeks post-op), Any Wound Complications

Primary Outcome Measure:

The primary outcome is the rate of contact allergic dermatitis or adverse skin reaction at 1 week post op and 1st post operative visit (2-3 weeks after surgery). We will also quantify time from surgery to reaction onset (Days). We will measure the size of the rash at post-operative follow up as well as classify the rash according to the classification system used in prior studies examining ACD.

Secondary Outcome Measures

1. Wound complications
2. Any workup for PJI (Serologic labs (ESR/CRP), arthrocentesis)
3. Any administration of post-operative antibiotics outside of normal protocol
4. Return to Operating Room for debridement, manipulation, other surgical interventions
5. Surgical Site Infection (SSI)
6. Confirmed Periprosthetic Joint Infection (PJI)
7. Stiffness requiring Manipulation Under Anesthesia (MUA)

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years that underwent primary total hip arthroplasty (THA)
2. Patients older than 18 years that underwent primary total or unicompartmental knee arthroplasty (TKA/UKA)

Exclusion Criteria:

1. Revision surgery
2. Prior history of allergic contact dermatitis
3. Prior history of non-TJA or UKA surgery with AQUACEL Ag dressing post-op
4. Occupational exposure to surgical dressings
5. Documented history of silver allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Rate of contact allergic dermatitis or adverse skin reaction at 1 week post surgery | 7 days post surgery
  Using a classification of skin reactions from mild, moderate to severe
Rate of contact allergic dermatitis or adverse skin reaction at 2-3 weeks post surgery | 2-3 weeks following surgery
  Using a classification of skin reactions from mild, moderate to severe

SECONDARY OUTCOMES:
Wound complications (if applicable) | 1 week post surgery
  If patients present with wound complications, require possible work up for infection, require antibiotics outside of normal protocol due to concerns of infection, return to the operating room, confirmed periprosthetic joint infection or stiffness that requires a manipulation under anesthesia
Wound complications (if applicable) | 2-3 weeks after surgery
  If patients present with wound complications, require possible work up for infection, require antibiotics outside of normal protocol due to concerns of infection, return to the operating room, confirmed periprosthetic joint infection or stiffness that requires a manipulation under anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Vasili Karas, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Once complete, we will share the summary of the data along with study protocol and SAP
Supporting Information: Study Protocol, SAP
Time Frame: Once the study is fully enrolled